CLINICAL TRIAL: NCT04123548
Title: A Multicenter, Open-label, Study of StrataGraft® Skin Tissue in Adult Subjects With Deep Partial-Thickness Thermal Burns
Brief Title: StrataGraft® Skin Tissue Expanded Access at Specific Study Sites ( StrataCAT )
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stratatech, a Mallinckrodt Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MNK01053115
Record Dates: First submitted 2019-10-06; First posted 2019-10-11 (Actual); Results first posted 2023-11-09 (Actual); Last update posted 2023-11-09 (Actual); Status verified 2023-10

CONDITIONS: Deep Partial-thickness Burn
Keywords: Alternative to Autograft

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- StrataGraft (Experimental): On Day 1, participants received a single application of up to 1:1 meshed StrataGraft skin tissue on up to 3 DPT wound(s) totaling no more than approximately 2000 square centimeters (cm^2) in area.
  Interventions: Biological: StrataGraft skin tissue

INTERVENTIONS:
Biological: StrataGraft skin tissue — StrataGraft skin tissue was delivered as a single topical application to no more than 3 separate burn sites, totaling up to approximately 2000 cm^2 of treatment area using no more than 20 tissues.
  Other Names: Experimental skin tissue

SUMMARY:
An autograft is a piece of skin taken from a healthy area of the body to be used to treat severe burns on another part of the same body.

StrataGraft skin tissue was an investigational tissue that could be used as an alternative to an autograft.

* StrataGraft skin tissue was in late-stage clinical development for the treatment of adults with deep partial-thickness (DPT) burns.
* There were no safety concerns reported to date. The sponsor submitted a treatment protocol to Food and Drug Administration (FDA) for doctors who participated in the Phase 3 Strata 2016 study (NCT 03005106) to allow for expanded access to StrataGraft before it was commercially available.

The main purpose of the study was to allow patients to receive StrataGraft during Biologics License Application review and prior to approval by the FDA for the treatment of DPT burns. The primary outcome measure was the number of participants with adverse events and safety concerns.

DETAILED DESCRIPTION:
The primary purpose of this trial was to provide expanded access to StrataGraft for thermally induced DPT burns that contained intact dermal elements and for which surgical excision and autograft would normally be part of the clinical management.

ELIGIBILITY:
Inclusion Criteria:

To be considered for inclusion, a participant must:

* Provide written informed consent
* Have enough healthy skin to reserve as donor site(s), in case autografting becomes necessary
* Have protocol-defined thermal burn(s) on the torso, upper extremities and lower extremities:

  1. that are the right size for treatment areas,
  2. with intact dermal elements for which excision and autografting are clinically indicated, and
  3. have not been previously excised and grafted.

Exclusion Criteria:

A participant must be excluded from participation if he/she:

* Is pregnant, a prisoner, or expected to live less than 3 months
* Has any other condition that, per protocol or in the opinion of the investigator, may compromise the participant's safety or the study objectives
* Has participated in an investigational study within 90 days before enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-01-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Stratatech, a Mallinckrodt Company
Locations (10):
- United States (10):
  - University of California Irvine, Orange, California
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - University of Florida (Health Shands Burn Center), Gainesville, Florida
  - University of Iowa, Iowa City, Iowa
  - Baton Rouge General, Baton Rouge, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - University of Missouri, Columbia, Missouri
  - Wake Forest University, Winston-Salem, North Carolina
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - University of Wisconsin Hospital, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Holmes Iv JH, Gibson ALF, Short T, Joe VC, Litt J, Carson J, Carter JE, Wibbenmeyer L, Hahn H, Smiell JM, Rutan R, Wu R, Shupp JW. A phase 3b, open-label, single-arm, multicenter, expanded-access study of the safety and clinical outcomes of StrataGraft(R) treatment in adults with deep partial-thickness thermal burns. Burns. 2024 Nov;50(8):2013-2022. doi: 10.1016/j.burns.2024.05.023. Epub 2024 Jun 6. PMID 39043513

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study across 10 study sites in the United States (US) from 21 February 2020 to 26 January 2022.
Pre-assignment Details: A total of 60 participants were screened of which, 52 participants were enrolled in the study.
Groups:
- StrataGraft: On Day 1, participants received a single application of up to 1:1 meshed StrataGraft skin tissue on up to 3 deep partial thickness (DPT) wound(s) totaling no more than approximately 2000 square centimeters (cm^2) in area.
Period: Overall Study
Arm/Group | StrataGraft
Started | 52
Completed | 38
Not Completed | 14
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 8
Not completed — Death | 4
Not completed — Reason Not Specified | 1

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (mITT) population included all participants who were enrolled and received StrataGraft.
Groups:
- StrataGraft: On Day 1, participants received a single application of up to 1:1 meshed StrataGraft skin tissue on up to 3 DPT wound(s) totaling no more than approximately 2000 cm^2 in area.
Arm/Group | StrataGraft
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.2 (17.00)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 50
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 42
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered casually related to the product.
  A TEAE is defined as an adverse event that started on or after the start of treatment (i.e. placement of StrataGraft).
Time Frame: AEs were collected on each individual participant for the duration of their study participation, i.e. from the time of signing the informed consent until study completion (up to approximately 7 months).
Population: mITT population included all participants who were enrolled and received StrataGraft.
Measure: Count of Participants; unit: Participants
Arm/Group | StrataGraft
Number analyzed (Participants) | 52
Participants | 46

ADVERSE EVENTS:
Time Frame: AEs were collected on each participant for the duration of the study participation i.e. from the time of signing the informed consent until study completion (up to approximately 7 months).
Description: mITT population included all participants who were enrolled and received StrataGraft. TEAEs are defined as those adverse events with onset date and time after the first placement of study product or those events in which the onset date and time are before the first placement of study product but worsened after the first placement of study product.
Arm/Group | StrataGraft
All-Cause Mortality (participants affected / at risk) | 4/52
Serious Adverse Events (participants affected / at risk) | 10/52
Other Adverse Events (participants affected / at risk) | 35/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | StrataGraft (N=52)
Arrhythmia (Cardiac disorders) | 1
Multiple organ dysfunction syndrome (General disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Intervertebral discitis (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Pneumonia staphylococcal (Infections and infestations) | 1
Septic shock (Infections and infestations) | 2
Wound infection (Infections and infestations) | 1
Intentional self-injury (Injury, poisoning and procedural complications) | 1
Tendon injury (Injury, poisoning and procedural complications) | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Nervous system disorder (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Myocardial infarction (Vascular disorders) | 1
Pulmonary embolism (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | StrataGraft (N=52)
Blood Loss anaemia (Blood and lymphatic system disorders) | 3
Constipation (Gastrointestinal disorders) | 5
Pain (General disorders) | 6
Neuralgia (Nervous system disorders) | 5
Delirium (Psychiatric disorders) | 3
Blister (Skin and subcutaneous tissue disorders) | 5
Cellulitis (Skin and subcutaneous tissue disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-10-02): https://cdn.clinicaltrials.gov/large-docs/48/NCT04123548/Prot_000.pdf
  • Statistical Analysis Plan (2022-03-11): https://cdn.clinicaltrials.gov/large-docs/48/NCT04123548/SAP_001.pdf